CLINICAL TRIAL: NCT00911339
Title: Mobilization of Endothelial Progenitor Cells Induced by Atorvastatin in Patients With Stable Coronary Artery Disease Treated With Anti-CD 34 Antibodies Coated Stents
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: prematurely interrupted because of difficulty in enrolment of patients.
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, FERRARIO, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Atorvastatin-CD34+
Record Dates: First submitted 2009-05-29; First posted 2009-06-01 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Stable Coronary Artery Disease
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin 10 mg (Active Comparator)
  Interventions: Drug: Atorvastatin
- Atorvastatin 80 mg (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 10 mg associated with stent genous
  Arms: Atorvastatin 10 mg
Drug: Atorvastatin — Atorvastatin 80 mg associated with stent genous
  Arms: Atorvastatin 80 mg

SUMMARY:
The purpose of this study is to evaluate the extent of the mobilization of endothelial progenitor cells induced by low versus high dose atorvastatin after 4 weeks of treatment, in patients treated with anti-CD 34 antibodies coated stent.

DETAILED DESCRIPTION:
Addition of statins to peripheral blood circulating mononuclear cells (PBMNCs) and to their CD 34+ subset cultures promotes endothelial progenitor cells (EPCs) proliferation, migration and survival according to a time and concentration-dependent effect. Data suggested that in patients with stable coronary artery disease atorvastatin 40 mg/day induced a 2 fold increase in the number of CD34+VEGFR2+ cells after 1 week of treatment and a 3 fold increase after 4 weeks; likewise, the number of EPCs colonies increased 1.5 times after 1 week and 3 times after 4 weeks. Data also suggested that the short term mobilizing effect of statins on EPCs may be transient and that medium-high doses long term statin treatment (> 1 month) may lead to a reduction in EPCs. Rather, a depletion of EPCs may not only be explained by exhausted mobilization but also by improved incorporation at sites of tissue hypoperfusion with potentially beneficial effects in therapeutic angiogenesis.In an interventional contest high concentrations of circulating EPCs may contribute to accelerate the reendothelialization process after stents implantation in coronary arteries. Considering the use of recent stents coated with anti-CD34 murine antibodies, the presence of high levels of PBMNCs expressing CD34 surface antigen may define the safety and efficacy levels of the procedure. Both the angiographic outcome and the clinical outcome seems to be better in patients with normal levels of EPCs than in patients with low levels. No data are available about the effects of different doses of statins on the biology of the PBMNCs and in particular about the timing of mobilization, duration of mobilization, the CD 34+ cell subset subpopulation mobilized and their gene expression balance in humans. No data are available about the effect of statins on clinical evolution in patients treated with PCI after the implantation of the stents coated by anti-CD34 murine antibodies.no specific data describing the effects of different doses of statins on the biology of the PBMNCs and in particular about the timing of mobilization, the duration of mobilization, the CD 34+ cell subset subpopulation mobilized and their gene expression balance in humans. No study has evaluated the effect of statins on clinical evolution in patients treated with PCI after the implantation of the new stents, coated by anti-CD34 murine antibodies. These data can contribute to better define the process of mobilization of endothelial progenitors induced by statins and to set up the best pharmacological strategy anti-CD34 coated stents deployment.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* stable angina or silent ischemia
* documented CAD
* signed written informed consent

Exclusion Criteria:

* current or recent therapy (stop < 3 months) with statins
* allergy to ASA or ticlopidine/clopidogrel
* myocardial infarction (< 3 months)
* recent significant trauma or surgical interventions (< 3 mesi)
* significant renal or hepatic diseases
* coagulative-hematological disorders
* cancer
* inflammatory diseases
* myopathy
* pregnancy (a pregnancy test will be performed in fertile women)
* severe coronary calcification, or small vessels disease (< 2.5 mm), long lesions (> 20 mm), ostial lesions, bifurcation lesions requesting treatment of the collateral vessel, multi-vessel disease requiring PCI before the completion of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
To evaluate the extent of the mobilization of endothelial progenitor cells induced by low versus high dose atorvastatin after 4 weeks of treatment, in patients treated with anti-CD 34 antibodies coated stent. | 7-28-90 days after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Irccs Policlinico San Matteo, Pavia, Italy